CLINICAL TRIAL: NCT00848250
Title: Effects of Angiotensin Converting Enzyme Inhibition During and After Cardiopulmonary Bypass in Infants and Children With Congenital Heart Defects
Brief Title: Angiotensin Converting Enzyme Inhibitors During Cardiopulmonary Bypass in Infants and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Gregory Fleming, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 071078
Record Dates: First submitted 2009-02-05; First posted 2009-02-20 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Congenital Heart Disease
Keywords: Cardiopulmonary Bypass; ACE inhibitor; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE inhibitor (Experimental): Patients already on an ACE inhibitor will continue it until the day of surgery
  Interventions: Drug: Angiotensin Converting Enzyme Inhibitor
- No ACE inhibitor (Experimental): Patients on ACE inhibitors who are randomized to stop their ACE inhibitor 48 hours prior to surgery
  Interventions: Other: No ACE Inhibitor

INTERVENTIONS:
Drug: Angiotensin Converting Enzyme Inhibitor — Patients randomized to this group will continue their current dose of ACE inhibitors until surgery
  Arms: ACE inhibitor
Other: No ACE Inhibitor — Patients randomized to this group will stop their ACE inhibitors 48 hours before surgery
  Arms: No ACE inhibitor

SUMMARY:
The purpose of this study is to determine whether ACE inhibitors alter the fibrinolytic, inflammatory, and hemodynamic response to cardiopulmonary bypass in infants and children with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Infants or children (newborn to 17 years of age) undergoing cardiopulmonary bypass for elective surgical correction of a congenital heart defect.
* Patients must be taking an ACE inhibitor prior to their operation

Exclusion Criteria:

* Patients in which discontinuing ACEIs is deemed unsafe by their primary cardiologist
* Any condition rendering the subjects legal guardian unable to understand the nature, scope, and possible consequences of the study.
* Pregnancy as ruled out by standard of care screening procedures.
* Individuals whose weight is less than 3.5 kg at the time of enrollment.
* Inability to comply with the protocol. ie. Children in whom it is deemed unsafe to have the extra blood draws, and children who are thought to be noncompliant with their medications.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fleming, MD, Principal Investigator — Vanderbilt University Medical Center, Division of Pediatric Cardiology; Mias Pretorius, MBChB, MSCI, Study Director — Vanderbilt University Medical Center, Department of Anesthesiology
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 participants were eligible, 8 refused participation
Period: Overall Study
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — surgery was completed without cardiopulm | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACE Inhibitor | No ACE Inhibitor | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.7 (3.5) | 20.8 (6.5) | 17.2 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: (PAI-1) Plasminogen Activator Inhibitor -1 Antigen
Time Frame: Baseline (prior to surgery), On CPB for 30 minutes, At completion of CPB, and postoperative day 1 (at 8:00AM)postoperative day 1
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- ACE Inhibitor; No ACE Inhibitor: Patients on ACE inhibitors who are randomized to stop their ACE inhibitor 48 hours prior to surgery
  No ACE Inhibitor: Patients randomized to this group will stop their ACE inhibitors 48 hours before surgery
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
ng/ml
  Baseline, Pre- Cardiopulmonary bypass (CPD) | 4.59 (2.36) | 3.78 (0.58)
  at 30 minutes on CPB | 13.59 (2.8) | 17.8 (2.49)
  Completion of CPB | 54.74 (6.63) | 58.56 (0.86)
  postoperative day 1 (at 8:00AM) | 57.13 (12.14) | 88.74 (14.02)
Statistical Analysis 1: Comparison: ACE Inhibitor vs No ACE Inhibitor; Test type: Superiority; p = 0.03, ANOVA

2. Primary Outcome: t-PA (Tissue-type Plasminogen Activator) Antigen
Time Frame: Baseline (prior to surgery) to postoperative day 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
ng/ml
  Baseline, Pre- Cardiopulmonary bypass (CPD) | 10.81 (1.0) | 8.31 (0.94)
  On CPB for 30 minutes | 12.97 (5.43) | 20.44 (6.38)
  At completion of CPB | 16.83 (1.84) | 28.03 (3.15)
  postoperative day 1 (at 8:00AM) | 14.36 (3.05) | 20.24 (1.82)
Statistical Analysis 1: Comparison: ACE Inhibitor vs No ACE Inhibitor; Test type: Superiority; p = 0.13, ANOVA; Repeated measures

3. Secondary Outcome: IL-6 (Interleukin-6)
Time Frame: Baseline (pre-surgery) to postoperative day 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
pg/ml
  Baseline, Pre- Cardiopulmonary bypass (CPD) | 2.29 (1.27) | 3.06 (1.76)
  on CPB for 30min | 9.64 (3.23) | 13.08 (3.49)
  At completion of CPB | 215.84 (32.59) | 141.00 (91.56)
  postoperative day 1 (at 8:00AM) | 401.69 (123.66) | 119.13 (33.54)
Statistical Analysis 1: Comparison: ACE Inhibitor vs No ACE Inhibitor; Test type: Superiority; p = 0.02, ANOVA; Repeated measures

4. Secondary Outcome: IL-8 (Interleukin-8)
Time Frame: Baseline (pre-surgery) to postoperative day 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
pg/mL
  Baseline (Before going on cardiopulmonary bypass | 11.69 (2.07) | 15.56 (3.61)
  at 30 minutes on CPB | 20.76 (4.57) | 36.91 (16.92)
  Admission to ICU following surgery | 213.74 (39.39) | 244.86 (121.13)
  postoperative day 1 (at 8:00AM) | 201.05 (66.91) | 127.03 (42.48)
Statistical Analysis 1: Comparison: ACE Inhibitor vs No ACE Inhibitor; Test type: Superiority; p = 0.67, ANOVA; Repeated measures

5. Secondary Outcome: (MAP) Mean Arterial Blood Pressure
Time Frame: Baseline (prior to surgery) to postoperative day 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
mmHg
  Baseline, Pre- Cardiopulmonary bypass (CPD) | 42.65 (1.68) | 47.82 (3.6)
  at 30 minutes on CPB | 53.02 (3.16) | 53.52 (2.93)
  At completion of CPB | 60.35 (4.23) | 59.48 (3.81)
  postoperative day 1 (at 8:00AM) | 60.63 (4.23) | 64.16 (3.33)

6. Secondary Outcome: Postoperative Bleeding
Description: Chest tube output at 4 and 24 hours after completion of surgery
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: mL/kg
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
mL/kg
  Chest tube output in 4 hrs | 38.4 (13.8) | 19.8 (2.9)
  Chest tube output in 24 hrs | 76.3 (20.7) | 43.2 (6.2)
Statistical Analysis 1: Comparison: ACE Inhibitor vs No ACE Inhibitor; P-value is for comparison of chest tube output at 24 hours; Test type: Superiority; p = 0.47, t-test, 2 sided

7. Secondary Outcome: Postoperative Renal Function
Description: Acute kidney injury occurring
Time Frame: Baseline (prior to surgery) to postoperative day 1
Measure: Number; unit: Percentage of subject with AKI
Arm/Group | ACE Inhibitor | No ACE Inhibitor
Number analyzed (Participants) | 11 | 9
Percentage of subject with AKI | 54.5 | 33.3
Statistical Analysis 1: Comparison: ACE Inhibitor vs No ACE Inhibitor; Test type: Superiority; p = 0.41, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the start of surgery until hospital discharge, approximately 7 days
Arm/Group | ACE Inhibitor | No ACE Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/11 | 2/9
Other Adverse Events (participants affected / at risk) | 4/11 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE Inhibitor (N=11) | No ACE Inhibitor (N=9)
ECMO (Cardiac disorders) | 1 (1) | 0 (0) — Extracorporeal membrane oxygenation
Surgical re-exploration (Surgical and medical procedures) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE Inhibitor (N=11) | No ACE Inhibitor (N=9)
Permanent pacemaker (Cardiac disorders) | 1 (1) | 0 (0) — Did the patient require a permanent pacemaker after surgery?
Pleural effusion (Cardiac disorders) | 3 (3) | 0 (0) — Did the patient develop a pleural effusion?

LIMITATIONS AND CAVEATS:
While patients were randomized to preoperative ACE inhibition, the present study was neither blinded nor placebo-controlled. However, the dose and type of ACE inhibitor were similar between the two study groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No